CLINICAL TRIAL: NCT05224167
Title: Melatonin Versus Hydroxizin for Pre Operative Anxiety in Elderly Patients With Hip Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, Professor head of anesthesia and intensive care department, Mongi Slim Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Melatonin versus Hydroxizin
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Preoperative Anxiety
Keywords: Melatonin; Hydroxizin; Hip fracture
MeSH Terms: conditions — Hip Fractures | interventions — Melatonin; Administration, Sublingual; Hydroxyzine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): patients of this group will receive 5 mg of Melatonin 12 hours and 5 mg 2 hours prior to surgery
  Interventions: Drug: Melatonin 5 MG Sublingual Tablet
- Group B (Active Comparator): patients of this group will receive 1 mg/kg of Hydroxizin 12 hours and 1 mg/ kg 2 hours prior to surgery
  Interventions: Drug: Hydroxyzine

INTERVENTIONS:
Drug: Melatonin 5 MG Sublingual Tablet — Melatonin 5 mg 12 hours and 2 hours prior to surgery
  Arms: Group A
Drug: Hydroxyzine — Hydroxyzine 1mg/kg 12 hours and 2 hours prior to surgery
  Arms: Group B

SUMMARY:
prospective randomized trial including adukt patients scheduled for hip fracture surgery, Randomization into 2 groups: Group A: Hydroxizin peroperatively Group B: Melatonin pre operatively

DETAILED DESCRIPTION:
prospective randomized trial including adukt patients scheduled for hip fracture surgery, Randomization into 2 groups: Group A: Hydroxizin peroperatively Group B: Melatonin pre operatively

Non inclusion criteria: patients with severe cognitive impairement Primary outcome pre operative anxiety assessed with Amsterdam preoperative anxiety and information scale

ELIGIBILITY:
Inclusion Criteria:

* All adult patients scheduled for hip fracture surgery

Exclusion Criteria:

* Patients with contraindications for hydroxizine or Melatonin Patients with severe cognitive impairement

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
preoperative anxiety | 1 hour before surgery
  preoperative anxiety scale

IPD SHARING:
Plan to Share IPD: No